CLINICAL TRIAL: NCT07066371
Title: The Effect of Emotional Freedom Technique on Anxiety Levels in Patients Receiving Preventive Foot Wound Care and Treatment in the Postoperative Period
Brief Title: The Effect of Emotional Freedom Technique on Patients Receiving Preventive Foot Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan 10
Record Dates: First submitted 2025-04-03; First posted 2025-07-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Limb Injury; Limb Ischemia; Complication Diabetic; Complication,Postoperative; Compliance, Patient; Anxiety
Keywords: post-operative; emotional freedom technique; anxiety; wound care
MeSH Terms: conditions — Diabetes Complications; Postoperative Complications; Patient Compliance; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pretestpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional freedom technique (Experimental): After the patients are given EFT training, they will be asked to apply it twice a week for 1 month. EFT videos and brochures will be given to the patients. 1 EFT session is applied for an average of 15 minutes.
  Emotional Freedom Technique Application Guidelines
  1. Determination of Subjective Units of Disturbance (SUD)
  2. Preparation or setup
  3. Application of appropriate acupuncture points in order
  4. 9-Gamut: An application that allows the two hemispheres of the brain to be stimulated simultaneously
  5. Application of appropriate acupuncture points in order again
  6. Control of the differentiation in the level of discomfort with SUDS again
  Interventions: Behavioral: Emotional freedom technique
- Standard of Care (No Intervention): As part of the pre-test, the patient introduction form, state and trait anxiety scale will be applied to the control group patients. The intervention will not be applied to the control group patients and the clinic's routine patient care and practices will continue. As part of the post-test, the state and trait anxiety scale will be applied to the control group patients again.
  *After the data collection process is completed, EFT training will be provided to the control group patients upon their request. EFT videos and brochures will be provided to the patients. It will be stated to the patients that they can contact the researchers by phone for information/support regarding the practices.

INTERVENTIONS:
Behavioral: Emotional freedom technique — Emotional Freedom Technique Application Guidelines
  1. Determination of Subjective Units of Disturbance (SUD)
  2. Preparation or setup
  3. Application of appropriate acupuncture points in order
  4. 9-Gamut: An application that allows the two hemispheres of the brain to be stimulated simultaneously
  5. Application of appropriate acupuncture points in order again
  6. Control of the differentiation in the level of discomfort with SUDS again
  Arms: Emotional freedom technique

SUMMARY:
It is planned to examine the effect of the emotional liberation technique on the anxiety level in patients who receive preventive foot wound care and treatment in the postoperative period.

H0: The emotional liberation technique has no effect on the anxiety level in patients who receive preventive foot wound care and treatment in the postoperative period.

H1: The emotional liberation technique has an effect on reducing anxiety in patients who receive preventive foot wound care and treatment in the postoperative period.

DETAILED DESCRIPTION:
The type of the study is a prospective randomized controlled clinical research model. The study design is a pre-test-post-test control group experimental trial. Data will be collected by the researchers through face-to-face interviews.

Patient identification form, state and trait anxiety scale will be applied to the experimental and control group patients as part of the pre-test. After the patients are given EFT training, they will be asked to apply it twice a week for 1 month. EFT videos and brochures will be given to the patients. 1 EFT session is applied for an average of 15 minutes. No intervention will be applied to the control group patients and the clinic's routine patient care and applications will be continued. State and trait anxiety scale will be applied to the experimental and control group patients as part of the post-test.

*After the data collection process is completed, EFT training will be given to the control group patients if they wish. EFT videos and brochures will be given to the patients. It will be stated to the patients that they can contact the researchers by phone for information/support regarding the applications.

Emotional freedom technique application is an application that works on cognitive and energetic levels. For this reason, in the application of the emotional freedom technique, exposure therapy is applied to individuals first. Exposure therapy is the comparison of individuals with the situation called trigger, which creates a stress response in the individual, during the application. The individual is reminded of the trigger and the individual is made conscious and aware of the discomfort. This situation activates the amygdala and creates a threat warning.

Emotional Freedom Technique Application Guidelines

1. Determination of Subjective Units of Disturbance (SUD)
2. Preparation or setup
3. Application of appropriate acupuncture points in order
4. 9-Gamut: An application that allows the two hemispheres of the brain to be stimulated simultaneously
5. Application of appropriate acupuncture points in order again
6. Control of the differentiation in the level of discomfort with SUDS again

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or older
* Must have no communication problems
* Must have had surgery for a foot ulcer

Exclusion Criteria:

* Having any auditory or mental problems
* Having difficulty/not being able to apply Emotional Freedom Technique (EFT)
* Wanting to leave the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
anxiety level | After receiving EFT training, patients will be asked to apply it twice a week for one month. Each EFT session lasts approximately 15 minutes. Measurements will be taken over one month.
  State and Trait Anxiety Scale:
  The adaptation and arrangement of the scales to Turkish was made by Necla Öner and Le Compte. Both scales consist of 20 items and are graded on a 4-point Likert scale. Scoring is done between 1-4. The scores obtained from both scales theoretically vary between 20 and 80. A high score indicates a high level of anxiety, a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, PhD., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)